CLINICAL TRIAL: NCT04904939
Title: Endobronchial Mucosal Biopsy in Patients With Suspected Pulmonary Sarcoidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abdelhady, Dr. Ahmed Abdelhady, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0106187
Record Dates: First submitted 2021-05-23; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Endobronchial Mucosal Pathology in Pulmonary Sarcoidosis
Keywords: Sarcoidosis - Bronchoscopy - Endobronchial biopsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The pathologist was blind to bronchoscopic mucosal changes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bronchoscopic mucosal biopsy — Endobronchial forceps biopsy using flexible bronchoscope

SUMMARY:
This prospective interventional study was done between May and September 2020. We included 20 patients from the chest department, Alexandria Main University Hospital (AMUH) with the inclusion criteria of having suspected pulmonary sarcoidosis (based on clinical and radiological presentation) and being ≥18 years of age. The bronchoscopy procedure was done under local anesthesia. Endobronchial biopsies and bronchoalveolar lavage were obtained.

DETAILED DESCRIPTION:
This prospective interventional study was done between May and September 2020. We included 20 patients from the chest department, Alexandria Main University Hospital (AMUH) with the inclusion criteria of having suspected pulmonary sarcoidosis (based on clinical and radiological presentation) and being ≥18 years of age. The patients who had any contraindication for flexible bronchoscopy (e.g. severe refractory hypoxemia, hemodynamic instability, uncorrectable bleeding diathesis, recent myocardial infarction or unstable angina) were excluded. The study was approved by the institutional ethics committee and an informed consent was taken from all patients before participation in the study according to the guidelines of ethics committee, Alexandria faculty of medicine.

All included patients were subjected to the followings: 1)full history taking including age, sex, history of other diseases and the presenting symptoms, 2)clinical examination including general examination and local chest examination, 3)routine laboratory investigations including complete blood picture, renal function tests, prothrombin activity and international normalized ratio (INR), 4)radiological evaluation including plain x-ray postero-anterior view and CT chest with IV contrast and 5) The bronchoscopy procedure that was performed by two experienced bronchoscopists.

The bronchoscopy procedure was done under local anesthesia with help of sedation by gradual doses of midazolam via the intravenous line. Any abnormal endoscopic findings suggestive of endobronchial sarcoidosis were reported by the operators. Bronchoalveolar lavage (BAL) was obtained by endoscopic injection of at least 120 cc of sterile saline then suction of the whole possible yield. Four endobronchial biopsies were obtained from the described findings plus two other biopsies from the main carina. In absence of mucosal abnormalities, four specimens were taken from a secondary carina and two were taken from the main carina. Immediate and 2 hours' postoperative clinical evaluation was done to detect any possible complications.

ELIGIBILITY:
Inclusion Criteria:

* Having suspected pulmonary sarcoidosis (based on clinical and radiological presentation) and being ≥18 years of age.

Exclusion Criteria:

* any contraindication for flexible bronchoscopy (e.g. severe refractory hypoxemia, hemodynamic instability, uncorrectable bleeding diathesis, recent myocardial infarction or unstable angina)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Pathological yield | 7 days
  Histopathological evidence of sarcoidosis in endobronchial mucosal biopsies

SECONDARY OUTCOMES:
Complications | 24 hours
  Bleeding, bronchospasm, fever, aspiration, pneumothorax, arrhythmia, hypoxia and cardiac arrest.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Abdelhady, Principal Investigator — Alexandria University
Locations (1):
- Alexandria Medicine Faculty, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
Study results

REFERENCES:
- [Background] Statement on sarcoidosis. Joint Statement of the American Thoracic Society (ATS), the European Respiratory Society (ERS) and the World Association of Sarcoidosis and Other Granulomatous Disorders (WASOG) adopted by the ATS Board of Directors and by the ERS Executive Committee, February 1999. Am J Respir Crit Care Med. 1999 Aug;160(2):736-55. doi: 10.1164/ajrccm.160.2.ats4-99. No abstract available. PMID 10430755
- [Background] Abdelhamid MA, Diab HS. The arrhythmic burden in patients with sarcoidosis. Is it a real concern? Egyptian Journal of Chest Diseases and Tuberculosis. 2016;65(1):311-7.
- [Background] Prasse A, Katic C, Germann M, Buchwald A, Zissel G, Muller-Quernheim J. Phenotyping sarcoidosis from a pulmonary perspective. Am J Respir Crit Care Med. 2008 Feb 1;177(3):330-6. doi: 10.1164/rccm.200705-742OC. Epub 2007 Nov 1. PMID 17975200
- [Background] Baughman RP, Winget DB, Bowen EH, Lower EE. Predicting respiratory failure in sarcoidosis patients. Sarcoidosis Vasc Diffuse Lung Dis. 1997 Sep;14(2):154-8. PMID 9306506
- [Background] Swigris JJ, Olson AL, Huie TJ, Fernandez-Perez ER, Solomon J, Sprunger D, Brown KK. Sarcoidosis-related mortality in the United States from 1988 to 2007. Am J Respir Crit Care Med. 2011 Jun 1;183(11):1524-30. doi: 10.1164/rccm.201010-1679OC. Epub 2011 Feb 17. PMID 21330454
- [Background] Baughman RP, Nunes H, Sweiss NJ, Lower EE. Established and experimental medical therapy of pulmonary sarcoidosis. Eur Respir J. 2013 Jun;41(6):1424-38. doi: 10.1183/09031936.00060612. Epub 2013 Feb 8. PMID 23397302
- [Background] Mason RJ, Broaddus VC, Martin TR, King TE, Schraufnagel D, Murray JF, et al. Murray and Nadel's Textbook of Respiratory Medicine E-Book: 2-Volume Set: Elsevier Health Sciences; 2010.
- [Background] Judson MA. The diagnosis of sarcoidosis. Clin Chest Med. 2008 Sep;29(3):415-27, viii. doi: 10.1016/j.ccm.2008.03.009. PMID 18539235
- [Background] Torrington KG, Shorr AF, Parker JW. Endobronchial disease and racial differences in pulmonary sarcoidosis. Chest. 1997 Mar;111(3):619-22. doi: 10.1378/chest.111.3.619. PMID 9118697
- [Background] Agarwal R, Srinivasan A, Aggarwal AN, Gupta D. Efficacy and safety of convex probe EBUS-TBNA in sarcoidosis: a systematic review and meta-analysis. Respir Med. 2012 Jun;106(6):883-92. doi: 10.1016/j.rmed.2012.02.014. Epub 2012 Mar 13. PMID 22417738
- [Background] Hewidy AA, Shebl AM. Efficacy and safety of bronchoscopic diagnostic procedures of sarcoidosis: a retrospective study. Egyptian Journal of Chest Diseases and Tuberculosis. 2016;65(2):473-8.